CLINICAL TRIAL: NCT01315912
Title: Dosage Optimization for Letrozole Treatment in Clomiphene Resistant Patients With Polycystic Ovary Syndrome: A Prospective Interventional Study
Brief Title: Dosage Optimization for Letrozole Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bushehr University of Medical Science (Other)
Responsible Party: Bushehr university of medical science, Bushehr university of medical science
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: bpums; bpums (Other: bpums)
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2008-01

CONDITIONS: Infertility
Keywords: clomiphene citrate; infertility; letrozole
MeSH Terms: conditions — Infertility | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Letrozole — 2.5 mg /day for 5 days
  Other Names: Femara

SUMMARY:
In a prospective interventional study, 44 Clomiphene resistant infertile patients were selected from Abolfazl Infertility Clinic of Bushehr University of Medical Sciences. Letrozole was given orally in a dose of 2.5mg, 5mg and 7.5mg, respectively. If the patient displayed no response, the dosage was increased. The size of follicle, endometrial thickness, estradiol, complications and clinical pregnancy rate were evaluated as the final outcome.

DETAILED DESCRIPTION:
In this prospective intervention, the investigators studied Abolfazle outpatients who were referred to us by Bushehr University of Medical Sciences in Iran between January 1, 2008 and December 30, 2010. The study was approved by the institutional Ethics Committee of Bushehr University of Medical Sciences and all patients were required to provide written informed consent before the study commenced.There were 3 steps in which the investigators prescribed letrozole (Femara,Novartis,Quebec,Canada). In all cases, daily administration began on the 3rd day of the menstrual cycle through to the 7th day (totaling 5 days). In the first step the investigators prescribed letrozole at a dose of 2.5 mg (one tablet) for one or two cycles according to the patient's response. Normal follicular size and endometrial thickness were considered 18-24 mm and 6 mm or more respectively.1 If the follicle was deemed not acceptable, the dose of letrozole was increased at the next cycle.

At the second and third steps the investigators prescribed letrozole at a dose of 5 mg daily and 7.5 mg/day,respectively and according to patient's response, repeat the same dose.

In the current study the investigators tested the hypothesis that prescribing letrozole as an ovulation induction agent in infertile women would increase pregnancy rate, ovulation and follicle number (at the normal size range of 18-24 mm), endometrial thickness (to normal thickness of 6 mm) and not have considerable side effects in the patients. The primary outcome measure was normal follicular size and the secondary outcome measure were the clinical and current pregnancy rates. Clinical pregnancy was considered as the presence of a gestational sac with fetal heart activity. Letrozole tablets were prescribed by an experienced nurse who throughly explained the method of use to the patients. Sonography was done by an experienced radiologist.

The nurse prescribed letrozole to the patients and the university hospital laboratory's technician did not know past medical history of clomiphene resistance of the patients. The radiologist did not have any knowledge about the drugs prescribed to the patients. Side effects and complications of Letrozole were detailed to all patients by an obstetrician. Statistical analysis was performed by the Statistical Package for Social Science version 11.5 for windows (SPSS Inc., Chicago. IL). The data was analyzed by student's t-test and chi-squared test for linear trend and comparing proportions. A P-value of <0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of polycystic ovarian syndrome(PCOS) patients diagnosed according to the Rotterdam criteria. The investigators defined Clomiphene citrate (Clomid, Iran hormone,Tehran,Iran) resistance as anovulation after consumption of 3 cycles of cc at 150 mg/day, determined by serial estradiol monitoring and sonography. Patients resistant to Clomiphene citrate became candidates for letrozole (Femara,Novartis,Quebec,Canada) consumption at the step-up of the protocol. Patients were between 18 and 39 years of age, body mass index (BMI) was > 19 or < 30 kg/m2 and day 3 follicle-stimulating hormone (FSH) < 12Miu/Ml.

Exclusion Criteria:

* abnormal thyroid Function test
* hyperprolactinoma
* galactorrhea
* male-factor infertility
* tubal and uterine causes of infertility (hysterosalpingography)
* abnormal response in progesterone challenge test which implies no endogenous estrogen production
* poor patient compliance
* complications with treatment

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
normal follicular size | two years

SECONDARY OUTCOMES:
clinical and current pregnancy rates | two years

CONTACTS AND LOCATIONS:
Overall Officials: Elham Rahmani, Dr, Principal Investigator — Bushehr University of Medical Science
Locations (1):
- Bushehr university of medical science, Bushehr, Bushehr, Iran

REFERENCES:
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742